CLINICAL TRIAL: NCT01249690
Title: Study of Efficacy of PAD-regimen(Bortezomib,Pirarubicin and Dexamethasone) and TAD-regimen(Thalidomide,Pirarubicin and Dexamethasone) in Newly Diagnosed Multiple Myeloma,Influence in Concentration of Bone Metabolites,and the Relations With Different Cytogenetic and Molecular Biological Changes
Brief Title: Efficacy Study of PAD and TAD in Newly Diagnosed Multiple Myeloma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Military Medical University (Other)
Collaborators: Zhejiang University (Other); Peking University People's Hospital (Other); Air Force Military Medical University, China (Other); Xiangya Hospital of Central South University (Other); Institute of Hematology & Blood Diseases Hospital, China (Other); Union hospital of Fujian Medical University (Other); Harbin Hematology and Oncology Institute (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Beijing Jishuitan Hospital (Other)
Responsible Party: Hou Jian/Director of department of hematology, Shanghai Changzheng Hospital, the Second Military Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHCZH-2010-CT-001
Record Dates: First submitted 2010-05-26; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-05

CONDITIONS: Multiple Myeloma
Keywords: Bortezomib,Thalidomide,bone metabolites
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PAD (Experimental)
  Interventions: Drug: Bortezomib,Pirarubicin,Dexamethasone
- TAD (Experimental)
  Interventions: Drug: Thalidomide,Pirarubicin,Dexamethasone

INTERVENTIONS:
Drug: Bortezomib,Pirarubicin,Dexamethasone — Bortezomib:1.3mg/m2,on day 1,4,8 and 11 of each 28 day cycle; Pirarubicin:10mg,on day 1 to 4 of each 28 day cycle; Dexamethasone:20mg,on day 1 to 4 and 8 to 11 of each 28 day cycle; Number of cycles: up to 8 cycles.
  Arms: PAD
Drug: Thalidomide,Pirarubicin,Dexamethasone — Thalidomide:200mg/d, everyday; Pirarubicin:10mg,on day 1 to 4 of each 28 day cycle; Dexamethasone:20mg,on day 1 to 4 and 8 to 11 of each 28 day cycle; Number of cycles: up to 8 cycles.
  Arms: TAD

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of PAD-regimen and TAD-regimen in newly diagnosed multiple myeloma(MM).

DETAILED DESCRIPTION:
Multiple myeloma (MM) is a malignant tumor with abnormal proliferation of monoclonal plasma cells in bone marrow. Bone damage is one of the characteristic clinical manifestations. Myeloma plasma cells and bone marrow microenvironment are the targets of thalidomide and bortezomib. The regimens based on them as first-line treatments of MM have greatly improved efficacy and prolonged the survival of MM patients. But whether the regimens can prevent and treat bone complications of MM patients or improve the quality of life is not clear. By evaluating the efficacy of PAD-regimen(Bortezomib,Pirarubicin and Dexamethasone) and TAD-regimen(Thalidomide,Pirarubicin and Dexamethasone) in MM and the effect of them on bone lesions, this study can provide evidence of evidence-based medicine for MM treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with symptomatic and measurable newly diagnosed Multiple Myeloma.
* Age > 18 years, KPS ≥ 60, and life expectancy of at least 3 months.
* Subjects must meet all of the following criteria within 14 days before starting therapy:

PLT≥50×109/L, Hb≥70 g/L, ANC≥0.75×109/L

* Subjects (or their legally acceptable representatives) must signed an informed consent document.

Exclusion Criteria:

* Severe cardiovascular disease ; HIV infection, or positive HBsAg, or active hepatitis C; HBV-DNA>104; hepatic functional parameter>2.5 times the upper limit of institutional laboratory normal.
* Grade 2 or more severe peripheral neuropathy or neuropathic pain; Grade 2 or more severe impaired hepatic and kidney function.
* Patient has radiotherapy or major surgery within 30 days before enrollment.
* Patient has hypersensitivity to boron, mannitol or thalidomide.
* Pregnant or breastfeeding women, or subject unwilling to use a method for contraception during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The overall response rate of PAD and TAD in patients with MM assessed by International Myeloma Working Group(IMWG) criteria | every treatment cycle

SECONDARY OUTCOMES:
The concentrations of bone metabolites | every two cycles
chromosome examination by cytogenetic and interphase Fluorescence in situ hybridization(FISH) method | at baseline
Overall survival(OS) and progression-free survival(FPS) | two and a half year
European Organisation for Research and Treatment of Cancer Quality Of life-Questionnaires-C30 (EORTC QLQ-C30) | every two cycles

CONTACTS AND LOCATIONS:
Overall Officials: Jian Hou, PhD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China